CLINICAL TRIAL: NCT00225173
Title: A Phase II Trial of Stanford VI ± Radiation Therapy in Locally Extensive and Advanced Stage Hodgkin's Disease With 3+ Risk Factors: the G6 Study
Brief Title: Combination Chemotherapy +/- Radiation in High Risk Hodgkin's Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G6HD; NIH/CA56060
Record Dates: First submitted 2005-09-21; First posted 2005-09-23 (Estimated); Last update posted 2014-08-27 (Estimated); Status verified 2005-09

CONDITIONS: Hodgkin Disease
Keywords: nodular sclerosis; lymphocyte rich; lymphocyte depleted; mixed cellularity
MeSH Terms: conditions — Hodgkin Disease | interventions — Doxorubicin; Vinblastine; Cyclophosphamide; Etoposide; etoposide phosphate; Vincristine; Bleomycin; Gemcitabine; Vinorelbine; Prednisone

ARMS (1):
- Treatment (Experimental): * Doxorubicin 25 mg/m2 IV w 1,3,5,7,9,11
  * Vinblastine 6 mg/m2 IV w 1,3,5,7,9,11
  * Cyclophosphamide 750 mg/m2 IV w 1, 5, 9
  * Etoposide2 60 mg/mg2 x 2 IV w 3, 7,11
  * Vincristine1 1.4 mg/m2 IV w 2,4,6,8,10,12 (cap @ 2mg)
  * Bleomycin 5 u/m2 IV w 2,4,6,8,10,12
  * Gemcitabine 1250 mg/m2 IV w 13,15,17,19
  * Vinorelbine 25 mg/m2 IV w 13,15,17,19
  * Prednisone 40 mg/m2 PO qod w 1-10, taper
  Interventions: Drug: Doxorubicin; Drug: Vinblastine; Drug: Cyclophosphamide; Drug: Etoposide; Drug: Vincristine; Drug: Bleomycin; Drug: Gemcitabine; Drug: Vinorelbine; Drug: Prednisone

INTERVENTIONS:
Drug: Doxorubicin — Doxorubicin 25 mg/m2 IV w 1,3,5,7,9,11
  Other Names: Adriamycin; hydroxydaunorubicin; hydroxydaunomycin
Drug: Vinblastine — Vinblastine 6 mg/m2 IV w 1,3,5,7,9,11
  Other Names: Alkaban-AQ; Velban; Vinblastine sulfate; Vincaleukoblastine; VLB
Drug: Cyclophosphamide — Cyclophosphamide 750 mg/m2 IV w 1, 5, 9
  Other Names: Cytoxan; Endoxan; Neosar; Procytox; Revimmune; cytophosphane
Drug: Etoposide — Etoposide2 60 mg/mg2 x 2 IV w 3, 7,11
  Other Names: Etopophos; Toposar; VePesid; etoposide phosphate; VP-16
Drug: Vincristine — Vincristine1 1.4 mg/m2 IV w 2,4,6,8,10,12 (cap @ 2mg)
  Other Names: Oncovin; leurocristine; VCR
Drug: Bleomycin — Bleomycin 5 u/m2 IV w 2,4,6,8,10,12
  Other Names: Blenoxane; bleomycin sulfate
Drug: Gemcitabine — Gemcitabine 1250 mg/m2 IV w 13,15,17,19
  Other Names: Gemzar; Gemcitabine HCl
Drug: Vinorelbine — Vinorelbine 25 mg/m2 IV w 13,15,17,19
  Other Names: Navelbine; Vinorelbine tartrate
Drug: Prednisone — Prednisone 40 mg/m2 PO qod w 1-10, taper
  Other Names: Deltasone; Liquid Pred

SUMMARY:
Patients with 3 or more adverse prognostic factors have a higher relapse rate. Significant anti-tumor activity in Hodgkin's lymphoma has been reported with two new drugs:gemcitabine and vinorelbine. The introduction of these new agents with their different mechanisms of action into the Stanford V regimen may increase effectiveness while maintaining a favorable toxicity profile with respect to fertility and a low risk of secondary leukemia. On this basis, we propose a new regimen, Stanford VI, for patients with bulky and advanced HD with 3 or more risk factors.

DETAILED DESCRIPTION:
Patients will receive chemotherapy weekly for 19 weeks, alone or followed by irradiation as indicated per protocol guidelines.

* Doxorubicin 25 mg/m2 IV w 1,3,5,7,9,11
* Vinblastine 6 mg/m2 IV w 1,3,5,7,9,11
* Cyclophosphamide 750 mg/m2 IV w 1, 5, 9
* Etoposide2 60 mg/mg2 x 2 IV w 3, 7,11
* Vincristine1 1.4 mg/m2 IV w 2,4,6,8,10,12 (cap @ 2mg)
* Bleomycin 5 u/m2 IV w 2,4,6,8,10,12
* Gemcitabine 1250 mg/m2 IV w 13,15,17,19
* Vinorelbine 25 mg/m2 IV w 13,15,17,19
* Prednisone 40 mg/m2 PO qod w 1-10, taper

ELIGIBILITY:
Inclusion Criteria:

* Untreated, locally extensive or advanced stage classical Hodgkin's disease
* 3 or more adverse risk factors
* Age > 18 years and < 70 years.
* No prior invasive malignancies for > 5 years except curatively-treated basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix.
* ECOG performance status 0 to 2
* WBC > 4000/µL
* Platelets > 100,000/µL
* Creatinine < 2.0mg/dL
* Bilirubin < 5.0mg/dL

Exclusion Criteria:

* HIV-positive
* Pregnant or currently breast feeding women
* Lymphocyte predominant Hodgkin's disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2001-10; Primary Completion 2005-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Freedom from progression

CONTACTS AND LOCATIONS:
Overall Officials: Sandra J. Horning, MD, Study Chair — Stanford University
Locations (1):
- Stanford University Medical Center, Stanford, California, United States